CLINICAL TRIAL: NCT04187716
Title: Multicenter Randomized Study on the Efficacy of Intravenous Iron Injection in Cancer Patients With Anemia
Brief Title: Intravenous Iron Injection in Cancer Patients With Anemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jun Ho Jang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-04-182-005
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Cancer Anaemia
MeSH Terms: interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferinject (Experimental): For patients undergoing chemotherapy, ferinject 1000mg will be injected within 24 hours or 24 hours after day 1 of the next chemotherapy cycle.
  Patients using targeted therapies can be dosed at any time after recognizing Hb 8.0-10.5g / dL and injecting 1000 mg of ferinject.
  Interventions: Drug: Ferinject
- remedies (Other): Treatment for anemia will include remedies such as iron (oral or intravenous), hematopoietic accelerators, and blood transfusions, and will be determined by researchers at each institution to provide optimal treatment for patients.
  Interventions: Drug: Ferinject

INTERVENTIONS:
Drug: Ferinject — For patients undergoing chemotherapy, ferinject 1000mg will be injected within 24 hours or 24 hours after day 1 of the next chemotherapy cycle.
  Patients using targeted therapies can be dosed at any time after recognizing Hb 8.0-10.5g / dL and injecting 1000 mg of ferinject.

SUMMARY:
* Multifactorial pathogenesis is involved in anemia of cancer patients and defining the causes of anemia is not always simple.
* Currently, treatment options available for anemia in cancer patients include red blood cell (RBC) transfusion, erythropoietin stimulating agent (ESA), and iron supplementation, accompanying considerable pros and cons for each treatment.
* Previous studies have demonstrated benefit when treating with IV iron in combination with ESA and, more recently, evidence is emerging to suggest a role for IV iron alone.
* In this study, investigator will assess the efficacy of intravenous iron for the treatment of anemia in cancer patients.
* Improvement of anemia and the improvement of quality of life compared to conservative treatment of intravenous iron

DETAILED DESCRIPTION:
This study is a comparative clinical trial of prospective, multicenter, randomized trials to evaluate the efficacy of intravenous iron (Ferinject®) in cancer patients with anemia.

Changes in hemoglobin in the treated and conservative treatment groups with a single intravenous Ferrinject® in patients with anemia by chemotherapy are identified.

1. Clinical Drug Ferinject Injection For patients undergoing chemotherapy, ferinject 1000mg will be injected within 24 hours or 24 hours after day 1 of the next chemotherapy cycle.

   Patients using targeted therapies can be dosed at any time after recognizing Hb 8.0-10.5g / dL and injecting 1000 mg of ferinject.
   * The administration of ferinject is a single dose, no re-administration. If chemotherapy is not performed, it can be administered at any time if the selection and exclusion criteria are met.
   * The administration period for ferinject should be administered within 24 hours or 24 hours after the day 1 of the chemotherapy cycle based on the results of phase 2 studies
2. remedies Within the period of sample collection of visits 2 to 4 after study enrollment, if the physician determines that treatment for clinically meaningful anemia is necessary, treatment for anemia other than ferinjects will be followed. Treatment for anemia will include remedies such as iron (oral or intravenous), hematopoietic accelerators, and blood transfusions, and will be determined by researchers at each institution to provide optimal treatment for patients. At the time this treatment is administered, the subject will be dropped from the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

The subject should be diagnosed with solid cancer or lymphoma. Hemoglobin level of test subject should be in the range of 8.0-10.5g / dL, or he / she has experienced hemoglobin reduction of 2g / dL or more during chemotherapy.

Exclusion Criteria:

The patients have a history of iron (oral or intravenous), hematopoietic stimulating agents (ESA), and dialysis within 4 weeks of study enrollment.

There is evidence that the patient's disease is a bone marrow invasion. There is a hypersensitivity reaction to ferinject or the components of ferinject.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The hemoglobin response is compared in patients treated with intravenous iron (Ferinject) and in conservatively treated patients. | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: JunHo Jang, ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea